CLINICAL TRIAL: NCT02706977
Title: The Effect of Dopamine on Diabetic Retinopathy
Acronym: Dopamine DR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Machelle Pardue, Adjunct Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00083672
Record Dates: First submitted 2016-03-04; First posted 2016-03-11 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Diabetes
Keywords: Ophthalmology
MeSH Terms: conditions — Diabetes Mellitus | interventions — carbidopa, levodopa drug combination; Electroretinography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Diabetes Group - Low Dose Sinemet CR (Experimental): Participants with diabetes mellitus type-2 and electroretinogram (ERG) delays will receive low dose Sinemet CR twice daily for two weeks.
  Interventions: Drug: Low Dose Sinemet CR; Device: RETeval Electroretinogram (ERG) Testing; Other: Contrast Sensitivity Testing; Other: Visual Acuity Testing
- Diabetes Group - High Dose Sinemet CR (Experimental): Participants with diabetes mellitus type-2 and electroretinogram (ERG) delays will receive high dose Sinemet CR twice daily for two weeks.
  Interventions: Drug: High Dose Sinemet CR; Device: RETeval Electroretinogram (ERG) Testing; Other: Contrast Sensitivity Testing; Other: Visual Acuity Testing
- Diabetes Group - No Electroretinogram (ERG) Delays (Other): Participants with diabetes mellitus type-2 who do not have electroretinogram (ERG) delays. Participants in this group will have one baseline visit only.
  Interventions: Device: RETeval Electroretinogram (ERG) Testing; Other: Contrast Sensitivity Testing; Other: Visual Acuity Testing
- Age-Matched Controls (Other): Participants will serve as age-matched controls for participants with diabetes. This group will participate in the baseline, week 2, and week 4 visits only.
  Interventions: Device: RETeval Electroretinogram (ERG) Testing; Other: Contrast Sensitivity Testing; Other: Visual Acuity Testing

INTERVENTIONS:
Drug: Low Dose Sinemet CR — Sinemet CR (25 mg carbidopa/100 mg levodopa) will be taken by mouth twice daily for two weeks.
  Arms: Diabetes Group - Low Dose Sinemet CR
Drug: High Dose Sinemet CR — Sinemet CR (50 mg carbidopa/200 mg levodopa) will be taken by mouth twice daily for two weeks.
  Arms: Diabetes Group - High Dose Sinemet CR
Device: RETeval Electroretinogram (ERG) Testing — ERG testing consists of sitting in the dark for 15 minutes. During the procedure, participants will have a single-use adhesive sensor strip placed on the skin near the eye. A hand-held device, called the RETeval, will be placed in front of the eye and a series of flashes and flickering lights presented. The light intensity level is typically not uncomfortable. When right eye imaging is complete, the procedure will be repeated on the left eye. Both eyes will be evaluated in less than 5 minutes for most participants. Electroretinogram (ERG) testing will be completed at baseline, day 1, week 2, and week 4.
Other: Contrast Sensitivity Testing — Contrast sensitivity testing consists of looking at a series of moving lines on a tablet device. The lines will change from white to grey to black. Participants will be asked to determine when they can no longer distinguish between the lines. Contrast sensitivity testing will be completed at baseline, day 1, week 2, and week 4.
Other: Visual Acuity Testing — Participants will be asked to look at an eye chart with letters or symbols that become smaller as they move from top to bottom of the chart. Visual acuity testing will be completed at baseline, day 1, week 2, and week 4.

SUMMARY:
The purpose of this study is to evaluate the use of electroretinogram (ERG) using a novel handheld system, RETeval, and evaluate contrast sensitivity testing in detecting pre-clinical retinopathy on a tablet device.

Investigators also seek to assess if a medication called Sinemet™ CR can improve the electrical functions of the eye in participants with diabetes mellitus. This study will include a total of 45 participants; 30 with diabetes mellitus and 15 age-matched non-diabetic controls. Participants with diabetes mellitus and electroretinogram (ERG) delays will be randomized to a low or high dose Sinemet CR group.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the use of electroretinogram (ERG) using a novel handheld system, RETeval, and evaluate contrast sensitivity testing in detecting pre-clinical retinopathy on a tablet device.

Investigators also seek to assess if a medication called Sinemet™ CR can improve the electrical functions of the eye in participants with diabetes mellitus. This study will include a total of 45 participants; 30 with diabetes mellitus and 15 age-matched non-diabetic controls. Participants with diabetes mellitus and electroretinogram (ERG) delays will be randomized to a low or high dose Sinemet™ CT group.

Age-matched controls will not receive Sinemet Ct drug treatment.

The study involves four visits over the course of 4 weeks, each visit consisting of 2-3 hours. Visual testing will be performed at 1 day and 2 weeks following treatment. The drug treatment will be halted and testing repeated again after a 2 week wash-out period.

ELIGIBILITY:
Inclusion Criteria

Participants with Diabetes Mellitus:

* Diagnosis of diabetes mellitus type-2
* HbA1c between 8 and 12%

Age-Matched Controls:

* Non-diabetic

Exclusion Criteria

Participants with Diabetes Mellitus:

* Currently taking dopamine-enhancing drugs (L-DOPA, bromocriptine)
* Currently taking nonselective monoamine oxidase (MAO) inhibitors
* Diagnosis of psychosis, Parkinson's disease, restless leg syndrome, major depression, confounding ocular disease (eg. visually significant cataract, glaucoma, macular degeneration, or retinitis pigmentosa)
* Pregnancy

Age-Matched Controls:

* Diabetes diagnosis
* Currently taking dopamine-enhancing drugs (L-DOPA, bromocriptine)
* Currently taking nonselective monoamine oxidase (MAO) inhibitors
* Diagnosis of psychosis, Parkinson's disease, restless leg syndrome, major depression, confounding ocular disease (eg. visually significant cataract, glaucoma, macular degeneration, or retinitis pigmentosa)
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Retinal Function assessed by Electroretinogram (ERG) Device | Baseline, Week 4
  The RETeval device consists of a hand-held wand with a pupil tracker. A skin electrode placed below the eye or DTL fiber records the response to flash stimuli. The pupil tracker provides feedback to the system so that the flash stimuli can compensate for the pupil size and produce the proper illumination to the retina. RETeval is intended to generate photopic signals and measure and display the electrical response signals generated by the retina and the visual nervous system using flash stimuli.
Change in Contrast Sensitivity assessed by the Contrast Sensitivity Function v1.0 (CSF v1.0) Tablet Application | Baseline, Week 4
  Participants will view the screen monocularly while wearing their normal correction. A drifting grating will be presented at 60 cm for 3, 6, 12 and 18 c/d. Following photopic testing (100 lux), the participant will be dark-adapted and a neutral density filter will be applied to the tablet screen to produce luminance of ~1 lux.
Change in Contrast Sensitivity assessed by the Sine Wave Grafting Test (CSV-1000E) | Baseline, Week 4
  The CSV-1000E is self-illuminated (85 cd/m2). A drifting grating will be presented at 60 cm for 3, 6, 12 and 18 c/d. The participant will view the chart from 2.5m. The intensity of the CSV-1000 will be reduced to 1 lux with neutral density filters for scotopic testing.
Change in Visual Acuity assessed by the Standard Snellen Static Chart | Baseline, Week 4
  The common Snellen chart is printed with eleven lines of block letters. The first line consists of one very large letter, which may be one of several letters, for example E, H, or N. Subsequent rows have increasing numbers of letters that decrease in size. Participants will cover one eye from 6 metres or 20 feet away, and read aloud the letters of each row, beginning at the top. The smallest row that can be read accurately indicates the visual acuity in that specific eye. The test will be repeated covering the opposite eye.

CONTACTS AND LOCATIONS:
Overall Officials: Machelle Pardue, PhD, Principal Investigator — Emory University
Locations (1):
- Atlanta VA Medical Center, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Motz CT, Chesler KC, Allen RS, Bales KL, Mees LM, Feola AJ, Maa AY, Olson DE, Thule PM, Iuvone PM, Hendrick AM, Pardue MT. Novel Detection and Restorative Levodopa Treatment for Preclinical Diabetic Retinopathy. Diabetes. 2020 Jul;69(7):1518-1527. doi: 10.2337/db19-0869. Epub 2020 Feb 12. PMID 32051147